CLINICAL TRIAL: NCT05741125
Title: Improving Appetite Self-Regulation in African American Adults With Type 2 Diabetes: A Digital Intervention
Brief Title: Improving Appetite Self-Regulation in African American Adults With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-2237
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; Binge Eating
Keywords: Bing Eating; Type 2 Diabetes; African Americans; Digital
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSMES + ASE intervention Appetite Self-Regulation (Centering Appetite) (Experimental): The Diabetes Self-Management Education and Support (DSMES) + Appetite Self-Regulation (ASE) intervention includes two, 45-60-minute group sessions delivered via telehealth. These sessions will enable participants to relearn their stomach's hunger and fullness signals and monitor their appetite. Participants will also learn strategies for glucose monitoring and carbohydrate management. Monthly booster sessions will be devoted to problem-solving, addressing barriers to emotion management, and self-monitoring type 2 diabetes mellitus symptoms. Participants will also receive weekly lessons with interactive activities delivered via a digital app.
  Interventions: Behavioral: DSME + ASE intervention (Centering Appetite)
- Control (No Intervention): Control group participants will attend two remotely delivered DSMES sessions that will offer content commonly. They will also receive weekly emails providing content from the American Association of Diabetes Educators.

INTERVENTIONS:
Behavioral: DSME + ASE intervention (Centering Appetite) — The intervention will enable participants to relearn their stomach's hunger and fullness signals and monitor their appetite. Participants will also learn strategies for glucose monitoring and carbohydrate management. Monthly booster sessions will be devoted to problem-solving, addressing barriers to emotion management, and self-monitoring type 2 diabetes mellitus symptoms. Participants will also receive weekly lessons with interactive activities delivered via a digital app.
  Other Names: Improving Appetite Self-Regulation in African American Adults with Type 2 Diabetes
  Arms: DSMES + ASE intervention Appetite Self-Regulation (Centering Appetite)

SUMMARY:
The purpose of this 6-month randomized clinical trial is to examine the feasibility of recruitment, attendance, retention, program adherence, and satisfaction of a digital application designed, Centering Appetite to improve glucose scores (HbA1c) and binge eating in African American adults with type 2 diabetes. Intervention participants will receive type 2 diabetes education and web-based lessons on appetite self-regulation. Participants will also receive a Fitbit to monitor daily physical activity. The investigators will follow up with participants at six months.

DETAILED DESCRIPTION:
Using a randomized clinical trial design examine the feasibility and acceptability of a 6-month digital diabetes self-management education program plus an appetite self-regulation intervention for (n=60) African Americans (AA) with type 2 diabetes who report uncontrolled eating in North Carolina. Sixty AAs will be randomized to the Centering Appetite intervention or the control group. Over the 6 months, Centering Appetite participants will have two intervention sessions supplemented by monthly booster sessions and weekly messages related to the program. The control group will also receive two intervention sessions and weekly nutrition tutorials. The study will examine the following: recruitment feasibility, attendance/retention, treatment adherence, intervention, HbA1c, and binge eating.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible if they

* identify as a Non-Hispanic, AA
* are over 18 years of age
* have an A1c value > 7.5
* have a working Smartphone
* complete binge eating screening

Exclusion Criteria:

Individuals will be excluded if they:

* have major end-organ type 2 diabetes mellitus complications
* have a history of weight loss surgery
* are currently pregnant
* in substance use treatment or are involved in another weight reduction program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Recruitment): The Percentage of Participants Who Were Eligible and Enrolled in the Study at Baseline | Baseline
  The number of potential participants screened for study eligibility versus the number of persons who enrolled in the study.
Feasibility (Recruitment): The Percentage of Participants Who Were Eligible and Enrolled in the Study at Month 6 | Month 6
  The number of potential participants screened for study eligibility versus the number of persons who enrolled in the study.
Feasibility (Attendance): The Percentage of Participants who Enrolled and Attended Each Intervention Session | Month 6
  The number of potential participants who attended intervention sessions versus the number of persons who enrolled in the study and did not attend intervention sessions.
Feasibility (Retention): The Percentage of Participants Retained in the Study at Month 6 | Month 6
  Percentage of participants retained in the study following enrollment.
Feasibility (Treatment Adherence): The Percentage of Participants Who Adhered to Study Protocol | Month 6
  Percentage of participants who adheres to study protocol.
Acceptability (Satisfaction): The Percentage of Participants Who Were Satisfied with the Delivery and Content of the Intervention | Month 6
  Participant satisfaction will be measured using a self-report scale at month 6. The Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM). This is a 4-item scale with 1 being the lowest measure and 5 being the highest measure.

SECONDARY OUTCOMES:
Changes in HbA1C | Baseline, Month 6
  Participant HbA1C will be measured using a glycohemoglobin analyzer.
Changes in Weight | Baseline, Month 6
  Participant body weight will be measured by trained research staff using a calibrated digital scale.
Changes in Blood Pressures (Systolic and Diastolic pressure) | Baseline, Month 6
  Participant blood pressures will be measured by trained research staff using a calibrated sphygmomanometer.
Changes in Binge Eating Episodes | Baseline, Month 6
  Participant binge eating episodes will be measured using the Binge Eating Scale (BES). This is a 16-item psychological self-assessment tool used to assess the severity of binge eating behavior. Minimum values are: 0-17 which indicates non-binge eating, and the maximum values are anything greater than 27, which indicates severe binge eating.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Goode, PhD, MPH, LCSW, Principal Investigator — University of North Carolina at Chapel Hil
Locations (2):
- United States (2):
  - Rachel W. Goode, Kannapolis, North Carolina
  - UNC Nutrition Research Institute, Kannapolis, North Carolina

IPD SHARING:
Plan to Share IPD: No